CLINICAL TRIAL: NCT03002025
Title: A Double-blind, Placebo-controlled, Randomized, Single-ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Subcutaneous Injection of JNJ-64304500 in Healthy Japanese and Caucasian Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Subcutaneous Injection of JNJ-64304500 in Healthy Japanese and Caucasian Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108267; 64304500CRD1001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: JNJ-64304500 50 milligram (mg) or placebo (Experimental): Participants (Japanese) will receive single subcutaneous (SC) dose of JNJ-64304500 50 mg or placebo on Day 1.
  Interventions: Drug: JNJ-64304500; Drug: Placebo
- Cohort 2: JNJ-64304500 150 mg or placebo (Experimental): Participants (Japanese) will receive single SC dose of JNJ-64304500 150 mg or placebo on Day 1.
  Interventions: Drug: JNJ-64304500; Drug: Placebo
- Cohort 3: JNJ-64304500 400 mg or placebo (Experimental): Participants (Japanese) will receive single SC dose of JNJ-64304500 400 mg or placebo on Day 1.
  Interventions: Drug: JNJ-64304500; Drug: Placebo
- Cohort 4: JNJ-64304500 150 mg or placebo (Experimental): Participants (Caucasian) will receive single subcutaneous (SC) dose of JNJ-64304500 150 mg or placebo on Day 1.
  Interventions: Drug: JNJ-64304500; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64304500 — Participants will receive JNJ-64304500 as SC injection.
Drug: Placebo — Participants will receive matching placebo to JNJ-64304500 as SC injection.

SUMMARY:
The primary purpose of this study is to assess the safety, tolerability, and pharmacokinetics (PK) following single-dose subcutaneous (SC) injection of JNJ-64304500 in healthy Japanese male participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have signed an informed consent document prior to any study related procedures indicating that they understand the purpose of the study including the procedures required and are willing to participate in the study
* Participant must be willing and able to adhere to the study visit schedule, prohibitions and restrictions specified in the protocol, and other protocol requirements
* Participant must have a body weight in the range of 60 to 90 kilogram (kg), inclusive, and a body mass index (BMI) of 18 to 30 kilogram per square meter (kg/m^2)
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must be a non-smoker for at least 3 months prior to study enrollment

Exclusion Criteria:

* Participant has a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant has an active acute or chronic infection (including chronic recurrent or invasive candidiasis) or diagnosed latent infection
* Participant has or has had a serious infection (example, sepsis, pneumonia or pyelonephritis), or have been hospitalized or received intravenous (IV) antibiotics for a serious infection during the 2 months prior to screening
* Participant has ever had a nontuberculous mycobacterial infection or opportunistic infection (eg, cytomegalovirus, pneumocystosis, and aspergillosis) prior to screening
* Participant has a history of active granulomatous infection, including histoplasmosis or coccidioidomycosis prior to screening
* If participant has had a chest radiograph within 3 months before study drug administration radiograph that shows an abnormality suggestive of a malignancy or current active infection, including tuberculosis (TB)

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-09-09 (Actual); Study Completion 2017-09-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to End of Study (Day 112)

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Up to End of Study (Day 112)
  The Cmax is the maximum observed serum analyte concentration.
Time to Reach Maximum Observed Serum Concentration (Tmax) | Up to End of Study (Day 112)
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Elimination Half-Life (t1/2) | Up to End of Study (Day 112)
  Elimination half-life associated with the terminal slope Lambda (z) of the semi logarithmic drug concentration-time curve, calculated as 0.693/Lambda (z).
Apparent Volume of Distribution (Vd/F) | Up to End of Study (Day 112)
  The Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Apparent Total Clearance (CL/F) | Up to End of Study (Day 112)
  The CL/F is defined as Dose/AUC (0-infinity).
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Up to End of Study (Day 112)
  The AUC (0-last) is the area under the serum concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Up to End of Study (Day 112)
  The AUC (0-infinity) is the area under the serum concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the serum concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Antibodies to JNJ-64304500 | Up to End of Study (Day 112)
  Serum samples will be collected and screened for antibodies binding to JNJ-64304500 and the titer of confirmed positive samples will be reported.
Percentage of Natural Killer Group 2 Member D Receptor Occupancy (NKG2D RO) by JNJ-64304500 | Up to End of Study (Day 112)
  Percentage of NKG2D receptors on natural killer (NK) cells and cluster of differentiation 8 (CD8)+ T cells that are occupied by JNJ-64304500 will be analyzed using a validated flow cytometry assay.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Tokyo, Japan